CLINICAL TRIAL: NCT04597658
Title: The Effectiveness of Body Weight Supported Treadmill Training in Stroke Patients: Randomized Controlled Study
Brief Title: The Effectiveness of Body Weight Supported Treadmill Training in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Elif Tarihçi, Principal Investigator, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ITF, PMR
Record Dates: First submitted 2020-10-18; First posted 2020-10-22 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Stroke; Cerebrovascular Accident; Gait Disorders, Neurologic; Walking, Difficulty
MeSH Terms: conditions — Stroke; Gait Disorders, Neurologic; Mobility Limitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional rehabilitation (Active Comparator)
  Interventions: Behavioral: Conventional rehabilitation
- Body weightsupported treadmill training (Experimental)
  Interventions: Behavioral: Bodyweight supported treadmill training (BWSTT)

INTERVENTIONS:
Behavioral: Bodyweight supported treadmill training (BWSTT) — In the BWSTT group, walking training will be given by asking the patients to walk on the treadmill as fast as they can, without exceeding the medium intensity according to the Borg scale. Bodyweight support will be gradually reduced according to the patient's tolerance.
  Arms: Body weightsupported treadmill training
Behavioral: Conventional rehabilitation — The conventional rehabilitation program includes posture and breathing exercises, lower extremity stretching, active-assistive range of motion and strengthening, balance-coordination exercises, and walking with a physiotherapist on a smooth surface.
  Arms: Conventional rehabilitation

SUMMARY:
In this study, the investigators aimed to evaluate the effects of exercise on body weight-supported treadmill in stroke patients on gait parameters, activity, body functions and quality of life, and to determine whether it has an effect on balance when applied in addition to conventional therapy.

DETAILED DESCRIPTION:
The study was planned as an open, prospective, randomized, single-blind study, and it was planned by the researchers to include 30 patients with stroke who applied to the Neurology outpatient clinic of Istanbul University, Istanbul Faculty of Medicine, Department of Physical Therapy and Rehabilitation. It was planned that the "Informed Consent Form" prepared before the study would be signed by the patient before being included in the study, and patient evaluation and follow-up forms would be filled in before and after the treatment.

Patients who meet the inclusion criteria at the beginning of the study will be numbered according to the order of application and randomly divided into two groups with the computer program. Group number 1 Treadmill with Weight Support; Group number 2 will be determined as the Conventional Rehabilitation group. In addition to the traditional rehabilitation program and rehabilitation program to both groups, one group will be given body weight support and treadmill therapy. The treatment will be applied as 15 sessions 5 days a week.

A traditional rehabilitation program will be applied to both groups. Posture and breathing exercises, lower extremity stretching, active auxiliary range of motion, and strengthening exercises will be applied. Electrical stimulation will not be delivered to the lower limb. Balance coordination exercises - sitting in a chair (individually shaped according to the patient's balance), holding it in a safe place if necessary; standing without support, standing quietly, heel tip, standing on one leg, and holding onto a chair). Patients will be asked to walk on a smooth surface in the company with a physiotherapist, using an assistive device, if any. The rehabilitation program is planned to last 30 minutes in total.

In the group where the bodyweight supported treadmill will be applied, patients will be asked to walk on the treadmill as fast as possible without exceeding the medium intensity according to the Borg scale. - Perceived fatigue on the Borg scale is quite mild 10-12. (40-50% of the maximum heart rate). Care should be taken that the patient wears appropriate shoes and clothing during walking.

In the beginning, 30% of the whole body weight will not be loaded. Bodyweight support will be reduced to 15% according to the tolerance of the patient. Later, when the patients can tolerate the speed of 2km / hour, they will not take more than two breaks during the 30-minute session, and 0% support will be applied when they are able to perform optimal walking without the need for at least 5 minutes of surveillance support. In the treatment to be performed under the guidance of a physiotherapist, manual intervention to the pelvis, trunk, and/or paretic extremity will correct the gait pattern. At the same time, verbal stimulation will ensure that temporal characteristics of the gait such as step length and walking speed are appropriate and at the same time the patient is motivated.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have had an ischemic or hemorrhagic stroke
* A history of the cerebrovascular event
* Patients who can walk 10 meters with or without an assistive device and / or orthosis (Patients with lower extremity motor functions above 2 according to Brunnstrom staging)
* Patients with comfortable walking speed <1.0 m / s
* Patients who can follow verbal warnings (patients with Mini-mental test score > 19)

Exclusion Criteria:

* Patients with a stroke less than a month
* Patients with stage 0 (non-functional ambulation) and stage 1 (the person's manual support is continuous) according to the functional ambulation scale
* Presence of serious cardiovascular or respiratory system diseases that prevent exercising
* Presence of uncontrolled metabolic disease (uncontrolled diabetes)
* Participation in an intensive rehabilitation program in the last month and continuing
* Presence of arthritis or severe contracture in the lower limb that may affect walking
* Presence of other accompanying neuromuscular diseases (such as Parkinson's disease)

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Change in The 10 Metre Walk Test | Baseline (before intervention), immediately after intervention
  The 10 Metre Walk Test is a performance measure used to assess walking speed in metres per second over a short distance.

SECONDARY OUTCOMES:
Change in The Rivermead Mobility Index Score | Baseline (before intervention), immediately after intervention
  The Rivermead Mobility Index is a one-dimensional index that focuses on measuring mobility status and includes basic mobility activities. It consists of 14 questions and one observation and includes a series of hierarchical activities from turning in bed to running.
Change in The 6 Minute Walk Test | Baseline (before intervention), immediately after intervention
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
Change in Stroke Specific Quality of Life Scale Score | Baseline (before intervention), immediately after intervention
  Stroke Specific Quality of Life Scale is one of the most comprehensive scales which measures quality of life in patients with stroke. It consists of 49 questions (each question is scored on a five points scale, 1-5) covering 12 domains (mobility, upper limb functions, social role, energy, self-care, family role, work-productivity, language, mood, personality, thinking, and vision). Each domain score is calculated by taking the unweighted means of associated questions while the unweighted mean of all the domains is used to calculate the total score.
Change in Tinetti Balance and Gait Assessment Score | Baseline (before intervention), immediately after intervention
  The Tinetti Assessment Tool is a simple, easily administered test that measures a resident's gait and balance. The test is scored on the resident's ability to perform specific tasks. Scoring of the Tinetti Assessment Tool is done on a three point ordinal scale with a range of 0 to 2. A score of 0 represents the most impairment, while a score of 2 represents independence. The individual scores are then combined to form three measures; an overall gait assessment score, and overall balance assessment score, ad a combined gait and balance score. The maximum score for the gait component is 12 points. The maximum score for the balance component is 16 points. The maximum total score is 28 points. IN general, residents who score below 19 are at a high risk for falls. Residents who score in the range of 19 - 24 points indicate that the resident has a risk for falls.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Tarihçi, MD, Principal Investigator — Istanbul University
Locations (1):
- Istanbul University Istanbul Faculty of Medicine, Department of Physical Medicine and Rehabilitation, Istanbul, Fatih, Turkey (Türkiye)

REFERENCES:
- [Background] Middleton A, Merlo-Rains A, Peters DM, Greene JV, Blanck EL, Moran R, Fritz SL. Body weight-supported treadmill training is no better than overground training for individuals with chronic stroke: a randomized controlled trial. Top Stroke Rehabil. 2014 Nov-Dec;21(6):462-76. doi: 10.1310/tsr2106-462. PMID 25467394
- [Background] Gama GL, Celestino ML, Barela JA, Forrester L, Whitall J, Barela AM. Effects of Gait Training With Body Weight Support on a Treadmill Versus Overground in Individuals With Stroke. Arch Phys Med Rehabil. 2017 Apr;98(4):738-745. doi: 10.1016/j.apmr.2016.11.022. Epub 2016 Dec 27. PMID 28034719
- [Background] Combs-Miller SA, Kalpathi Parameswaran A, Colburn D, Ertel T, Harmeyer A, Tucker L, Schmid AA. Body weight-supported treadmill training vs. overground walking training for persons with chronic stroke: a pilot randomized controlled trial. Clin Rehabil. 2014 Sep;28(9):873-84. doi: 10.1177/0269215514520773. Epub 2014 Feb 11. PMID 24519922
- [Derived] Tarihci Cakmak E, Yaliman A, Torna G, Sen EI. The effectiveness of bodyweight-supported treadmill training in stroke patients: randomized controlled trial. Neurol Sci. 2024 Jul;45(7):3277-3285. doi: 10.1007/s10072-024-07385-z. Epub 2024 Feb 16. PMID 38363446